CLINICAL TRIAL: NCT04103346
Title: Reducing Particulate Matter-associated Cardiovascular Health Effects for Seniors
Acronym: RAPIDS2-Ypsi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan State University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Geoffrey Barnes, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HUM00156608; 2R01NR014484-06 (NIH)
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cardiometabolic Health
MeSH Terms: interventions — Air Filters; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: crossover of active filtration in subject's residence with a home filtration unit (Holmes air filtration unit Model HAP8650B-NU-1) versus an inactive sham filtration
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: filtration units with or without filters. filters are placed by research assistant from the environmental college and researchers performing the health outcomes are blinded to the condition (sham or active filtration) along with the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- air filtration with hepa filter (Active Comparator): air purifier used is the Holmes HAP8650B-NU-1 with the hepa filter inserted.
  Interventions: Other: air filtration with air purifier with hepa filter
- air filtration with hepa filter removed (Sham Comparator): sham comparator uses the Holmes HAP8650B-NU-1 air purifier to be operated with the filter removed.
  Interventions: Other: sham

INTERVENTIONS:
Other: air filtration with air purifier with hepa filter — long-term (4 week) air filtration with the Holmes HAP8650B-NU-1 air purifier in the residence of low-income seniors impacted by roadway pollutants.
  Other Names: air filtration
  Arms: air filtration with hepa filter
Other: sham — air purifier running with air filter removed
  Other Names: air purifier running with air filter removed
  Arms: air filtration with hepa filter removed

SUMMARY:
Exposure to fine particulate matter (PM2.5) air pollution is an established risk factor for cardiovascular (CV) morbidity.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled (sham filtration) crossover trial comparing the effectiveness bedroom-only portable indoor air filtration units [AFUs] to reduce personal PM2.5 exposures and improve cardiometabolic health. The health benefits (primary outcome: resting BP) will be evaluated over acute (4-day) and long-term (4-week) periods in 50 nonsmoking elderly adults living in a senior facility impacted by near-roadway pollutants.

Because of COVID-19 restrictions that occurred during the trial, certain outcome measures were removed from the protocol, as they could not be performed: 24-hr Blood Pressure, Heart Rate Variability (HRV), BpTRU BP measurements, and WatchPAT. Other outcome measures were not removed from the protocol, but data could not be collected for them because of COVID restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker
* ≥60 years old
* residing in Carpenter Place Apartments

Exclusion Criteria:

* Active cigarette smoker
* daily secondhand smoke exposure (self-report)
* any CV event (myocardial infarction, stroke, heart failure, revascularization) in the past 3 months
* unstable CV condition or risk factor (uncontrolled diabetes, class 3-4 angina or heart failure) or any medical condition that would place the participant at risk from participation or jeopardize study integrity (per investigators)
* expected overnight travel outside their apartment during the 14-week study period
* unable to provide informed consent
* lung disease requiring oxygen
* renal dialysis
* cancer receiving active treatment or chemotherapy
* severe uncontrolled high BP ≥160/100 mm Hg or SBP<115 mm Hg.
* CV medication change in the prior month. If participants are on medications for high BP, diabetes, or a CV condition, they will need to have stable therapy during the prior month with no planned changes during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brook, MD, Principal Investigator — Wayne State University
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants withdrew from the trial prior to randomization. Of the 35 participants who were randomized, data from 2 was not included in the analyses, because of external factors that rendered the data from those participants unusable.
Groups:
- Air Filtration With Hepa Filter, Then With Hepa Filter Removed: air purifier used is the Holmes HAP8650B-NU-1 with the hepa filter inserted, then with the filter removed following washout (sham comparator).
  air filtration with air purifier with hepa filter: long-term (4 week) air filtration with the Holmes HAP8650B-NU-1 air purifier in the residence of low-income seniors impacted by roadway pollutants.
  sham: air purifier running with air filter removed
- Air Filtration Without Hepa Filter, Then With Hepa Filter: sham comparator used the Holmes HAP8650B-NU-1 air purifier to be operated without the filter, then with the hepa filter installed following washout.
  air filtration with air purifier with hepa filter: long-term (4 week) air filtration with the Holmes HAP8650B-NU-1 air purifier in the residence of low-income seniors impacted by roadway pollutants.
  sham: air purifier running with air filter removed
Period: Phase 1 - 4 Weeks
Arm/Group | Air Filtration With Hepa Filter, Then With Hepa Filter Removed | Air Filtration Without Hepa Filter, Then With Hepa Filter
Started | 21 | 12
Completed | 21 | 12
Not Completed | 0 | 0
Period: Washout - 2 Weeks
Arm/Group | Air Filtration With Hepa Filter, Then With Hepa Filter Removed | Air Filtration Without Hepa Filter, Then With Hepa Filter
Started | 21 | 12
Completed | 21 | 12
Not Completed | 0 | 0
Period: Phase II - 4 Weeks
Arm/Group | Air Filtration With Hepa Filter, Then With Hepa Filter Removed | Air Filtration Without Hepa Filter, Then With Hepa Filter
Started | 21 | 12
Completed | 21 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Filtration With Hepa Filter, Then With Hepa Filter Removed | Air Filtration Without Hepa Filter, Then With Hepa Filter | Total
Number analyzed (Participants) | 21 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.2 (7.11) | 72.5 (8.12) | 74.9 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 21 | 12 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 12 | 33
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.7 (6.21) | 30.2 (8.41) | 29.2 (6.99)
History of coronary artery disease [Count of Participants; unit: Participants]
  No | 15 | 8 | 23
  Yes | 6 | 4 | 10
History of cerebrovascular disease [Count of Participants; unit: Participants]
  No | 20 | 9 | 29
  Yes | 1 | 3 | 4
History of hyperlipidemia [Count of Participants; unit: Participants]
  No | 9 | 9 | 18
  Yes | 12 | 3 | 15
History of hypertension [Count of Participants; unit: Participants]
  No | 6 | 3 | 9
  Yes | 15 | 9 | 24
History of diabetes [Count of Participants; unit: Participants]
  No | 12 | 10 | 22
  Yes | 9 | 2 | 11
Blood Pressure Medication [Count of Participants; unit: Participants]
  No | 6 | 3 | 9
  Yes | 15 | 9 | 24
Statin [Count of Participants; unit: Participants]
  No | 9 | 9 | 18
  Yes | 12 | 3 | 15
Diabetes medication [Count of Participants; unit: Participants]
  No | 12 | 10 | 22
  Yes | 9 | 2 | 11
Aspirin [Count of Participants; unit: Participants]
  No | 14 | 8 | 22
  Yes | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure was measured twice a day, in the morning and the evening, from Tuesday through Friday during the first and fourth week of each of the four-week periods in which participants were exposed to one of the interventions. Results reflect the average of systolic readings taken.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 33 | 33
mm Hg | 127.0 (16.2) | 126.5 (16.0)
Statistical Analysis 1: Comparison: Air Filtration With Hepa Filter vs Air Filtration With Hepa Filter Removed; Test type: Superiority; p = 0.588, Mixed Effects Model

2. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure was measured twice a day, in the morning and the evening, from Tuesday through Friday during the first and fourth week of each of the four-week periods in which participants were exposed to one of the interventions. Results reflect the average of diastolic readings taken.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 33 | 33
mm Hg | 75.1 (10.6) | 75.3 (10.4)
Statistical Analysis 1: Comparison: Air Filtration With Hepa Filter vs Air Filtration With Hepa Filter Removed; Test type: Superiority; p = 0.748, Mixed Effects Model

3. Secondary Outcome: Atmospheric Particulate Matter (pm2.5) - Indoor
Description: Atmospheric particulate matter was measured daily in the units of ug/m3 and determined using a portable analyzer (PDR-1500). Results reflect the average amount of atmospheric particulate matter present per day.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: (µg/m3) per day
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 33 | 33
(µg/m3) per day | 1.3 (1.5) | 8.3 (12.8)
Statistical Analysis 1: Comparison: Air Filtration With Hepa Filter vs Air Filtration With Hepa Filter Removed; Test type: Superiority; p < 0.001, Mixed Effects Model

4. Secondary Outcome: Atmospheric Particulate Matter (pm2.5) - Outdoor
Description: Atmospheric particulate matter was measured daily in units of ug/m3 and determined using a portable analyzer (PDR-1500). Results reflect the average amount of atmospheric particulate matter present per day.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: (µg/m3) per day
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 33 | 33
(µg/m3) per day | 10.3 (5.8) | 8.9 (2.3)
Statistical Analysis 1: Comparison: Air Filtration With Hepa Filter vs Air Filtration With Hepa Filter Removed; Test type: Superiority; p = 0.0764, Mixed Effects Model

5. Secondary Outcome: 24-hr Personal PM2.5 (Filter-gravimetric Mass)
Description: PM2.5 mass measured from the filters contained in the personal particulate monitors worn for 24-hours by participants performed on the last week of each cross-over limb (twice per participant in total). 24-hour data collection for personal PM2.5 exposure was collected from Thursday morning at 9 am to Friday morning at 9 am during trial week 4 and during trial week 10.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: µg/m3 per 24-hour period
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 33 | 33
µg/m3 per 24-hour period | 5.1 (4.6) | 12.4 (15.6)
Statistical Analysis 1: Comparison: Air Filtration With Hepa Filter vs Air Filtration With Hepa Filter Removed; Test type: Superiority; p < 0.001, Mixed Effects Model

6. Secondary Outcome: Black Carbon, Hourly Personal PM2.5 Levels
Description: Evaluation of the effect of active vs sham filtration on lowering black carbon levels and hourly levels of PM2.5 throughout a 24-hour period.
Time Frame: 10 weeks
Population: This outcome was not performed because of COVID-19 restrictions in place during the trial, and no data for this outcome will be collected.
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Aortic Hemodynamics
Description: Determined using pulse wave analyses of the augmentation index calculated as the height of the reflected wave as a percentage of the total height of the ascending aortic pressure wave.
Time Frame: 10 weeks
Population: as for outcome 6
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Insulin Sensitivity
Description: To determine the impact of reduced particulate matter on insulin sensitivity, determined by measuring insulin and glucose to calculate the homeostasis model assessment of insulin resistance (HOMA-IR) metric.
Time Frame: 10 weeks
Population: as for outcome 6
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Adrenal Steroid Panel
Description: Panel of hair, saliva, blood
Time Frame: 10 weeks
Population: as for outcome 6
Arm/Group | Air Filtration With Hepa Filter | Air Filtration With Hepa Filter Removed
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Air Filtration Without Hepa Filter: sham comparator used the Holmes HAP8650B-NU-1 air purifier operated without the filter.
  sham: air purifier running with air filter removed
Arm/Group | Air Filtration With Hepa Filter | Air Filtration Without Hepa Filter
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT04103346/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04103346/ICF_001.pdf